CLINICAL TRIAL: NCT00202371
Title: Transfusion Effects in Myelodysplastic Patients: Limiting Exposure (Temple)
Brief Title: Transfusion Effects in Myelodysplastic Patients: Limiting Exposure
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Too few inclusions
Sponsor: Sanquin Research & Blood Bank Divisions (Other)
Collaborators: Ministry of Health, Welfare and Sports, The Netherlands (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-021
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2015-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS, Fatigue, RBC transfusion
MeSH Terms: conditions — Myelodysplastic Syndromes; Fatigue | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Red Blood Cell transfusion

SUMMARY:
The goal of this study was to compare a restrictive RBC transfusion policy (a Hb transfusion trigger: 7.2 gr/dl) with a more liberal RBC transfusion policy (a Hb transfusion trigger: 9.6 gr/dl) on physical fatigue.

DETAILED DESCRIPTION:
The goal of this study was to compare a restrictive RBC transfusion policy (a Hb transfusion trigger of 7.2 gr/dl) with a more liberal RBC transfusion policy (a Hb transfusion trigger of 9.6 gr/dl) on physical fatigue.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis myelodysplastic syndrome (primary or secondary) based on cytopenia in at least 1 cell line + dysplasia in 2 cell lines (and no other cause (especially deficiencies)) and a pathologic anatomic diagnosis after bone marrow punction.
* refractory anaemia (RA): blood: ≤ 1% blasts, ≤ 1 x 109 monocytes; bone marrow: < 5% blasts, ringed sideroblasts ≤ 15% of the erythroid cells
* refractory anaemia with ringed sideroblasts (RARS): blood: ≤ 1% blasts, ≤ 1 x 109 monocytes; bone marrow: < 5% blasts, ringed sideroblasts > 15% of the erythroid cells
* refractory anaemia with excess blasts (RAEB): blood: < 5% blasts, ≤ 1 x 109 monocytes; bone marrow: blasts ≥ 5 -≤ 20%
* chronic myelomonocytic leukaemia (CMML): blood: >1 x 109/l monocytes, <5% blasts; bone marrow: blasts < 20%, increase of the monocytic component
* erythrocyte transfusion need
* working knowledge of the national language
* written consent for participating this study (informed consent)

Exclusion Criteria:

* candidate for bone marrow- or organ transplantation
* medication: growth factors (GM-CSF), or EPO
* patients who will receive an intensive chemotherapeutic treatment with a cytopenia, expected longer than 2 weeks
* refractory anaemia with excess blasts in transformation (RAEB-t): blood: ≥ 5% blasts or Auer rods; bone marrow: or blasts > 20 - < 30% or Auer rods
* pregnancy at the moment of inclusion
* patients with congenital severe haemolytic anaemia, like thalassemia or sickle cell anaemia
* patients with AIDS or a severe congenital or acquired (e.g. iatrogenic) immunological disorder
* severe active infections at the moment of inclusion
* severe cardiac, pulmonal, neurological, metabolic or psychiatric disease at the moment of inclusion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-07; Study Completion 2005-07 (Estimated)

PRIMARY OUTCOMES:
fatigue

SECONDARY OUTCOMES:
Health related Quality of Life, Blood usage and the costs, Haemoglobin increase after transfusion, Heart beat, blood pressure, temperature, platelet count, Development of RBC alloantibodies, Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dick J van Rhenen, MD, PhD, Study Director — Sanquin Blood Bank South West Region
Locations (1):
- Sanquin Blood Bank South West Region, Rotterdam, Netherlands

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449